CLINICAL TRIAL: NCT05602402
Title: To Evaluate the Efficacy and Safety of CAEP-01 on Eye Strain in Children With Heavy Screen Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AP/220201/CAEP/ES
Record Dates: First submitted 2022-10-17; First posted 2022-11-02 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Vision Disorders
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Intervention Model Description: CAEP-01, Placebo Dose: 44 mg/day Route: orally for 84 ± 3 days Regimen: one capsule before breakfast (preferably with milk/butter/ghee)
Who Masked: Participant, Investigator
Masking Description: Sealed envelop, double-blind randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAEP-01 (Active Comparator): Dose: 1 capsule Route: orally for 84 ± 3 days Regimen: one capsule beforebreakfast (preferably with milk/butter/ghee)
  Interventions: Other: CAEP-01
- Placebo (Placebo Comparator): Dose: 1 capsule Route: orally for 84 ± 3 Regimen: one capsule before breakfast (preferably with milk/butter/ghee)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: CAEP-01 — Dose: 1 capsule Route: orally for 84 ± 3 days Regimen: one capsule before breakfast (preferably with milk/butter/ghee)
  Arms: CAEP-01
Other: Placebo — Dose: 1 capsule Route: orally for 84 ± 3 days Regimen: one capsule before breakfast (preferably with milk/butter/ghee)
  Arms: Placebo

SUMMARY:
Several recent clinical trials have highlighted the potential role of Product in promoting eye health.product whose structural and functional characteristics make it a promising bioactive compound in the prevention of several human diseases as well as in the maintenance of a good health status. it might relieve eyestrain in people using computer monitors as suggested who conducted a double-blind randomized clinical trial by enrolling visual display terminal workers and prescribed them product or placebo. Study outcomes were objectively evaluated by using a proper instrumentation to measure eye muscle endurance. Subjects receiving Product experienced a significant relief from eyestrain compared to the placebo group.

ELIGIBILITY:
Inclusion Criteria:

1. Girls and Boys between the ages 10 to 14.
2. Participants who have a history of using a digital device (phone, tablet, computer, etc) at least 4 hours per day, for minimum of last 3 months prior to screening.
3. Participants who have complained of eye strain on use of digital device.
4. Participant with CVS-Q score ≥ 8.
5. Participants who have history of playing video game for least 6 hours per week.
6. Best Corrected Visual Acuity (BCVA) of 20/20.
7. Participants with ≤ 12.5 cm and ≥ 6 cm amplitude on accommodation test.
8. Participants with parents who are literate enough to understand the essence of study, are informed about the purpose of the study, and understand their rights.
9. Participants with parents who are able to give written informed consent and willingness to participate in the study and comply with its procedures

Exclusion Criteria:

1. Participant with CVS-Q score ≥ 19.
2. Asthenopia Visual Fatigue Likert Scale Score ≤ 2 for each symptom.
3. Near Point Convergence (NPC) no further than 10 cm
4. Stereopsis of ≥ 40 arc/sec
5. Not diagnosed with amblyopia
6. Refractive error less than -3 or more than +2
7. Participants who wear contact lenses.
8. Participants with any diagnosed ocular motility disorder or accommodative/binocular vision issues.
9. Participants with a history of eye alignment or binocularity issues.
10. Participants who are color-blind.
11. Participant on any antioxidant, retinols and carotenoid supplements.
12. Participants who have used eye care products within 3 months prior to the screening visit.
13. Participants who have been diagnosed with Type I diabetes.
14. Participants who have been diagnosed with Covid-19 one month before the screening visit.
15. Participants scheduled to receive any vaccination during the study period.
16. Participants who have immunosuppressive disorders or are taking immunosuppressive medication.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-04-24 (Actual)

PRIMARY OUTCOMES:
Computer Vision Syndrome-Questionnaire | Screening before playing videogames on digital device
  To assess the effect of 84 days of IP consumption on severity of the symptoms using Computer Vision Syndrome-Questionnaire.The two levels of intensity, or strength of the symptom, will be graded similarly, on a scale of 1 to 2 points, where moderate = 1 and intense = 2. In the analysis, a symptom rated as never occurring will be treated as 0 (none) on the intensity scale.
  The overall assessment will be conducted by obtaining the total score for DES. The result of frequency X intensity will be recorded as: 0 = 0; 1 or 2 = 1; 4 = 2. If the total score is ≥ 6 points, the participant will be considered to be suffering from digital eye strain. It is further categorized as mild DES (score = 6-12), moderate DES (score = 13-18), and severe DES (score = 19-32)
Computer Vision Syndrome-Questionnaire | Day 0 before playing videogames on digital device
  To assess the effect of 84 days of IP consumption on severity of the symptoms using Computer Vision Syndrome-Questionnaire.The two levels of intensity, or strength of the symptom, will be graded similarly, on a scale of 1 to 2 points, where moderate = 1 and intense = 2. In the analysis, a symptom rated as never occurring will be treated as 0 (none) on the intensity scale.
  The overall assessment will be conducted by obtaining the total score for DES. The result of frequency X intensity will be recorded as: 0 = 0; 1 or 2 = 1; 4 = 2. If the total score is ≥ 6 points, the participant will be considered to be suffering from digital eye strain. It is further categorized as mild DES (score = 6-12), moderate DES (score = 13-18), and severe DES (score = 19-32)
Computer Vision Syndrome-Questionnaire | Day 14 before playing videogames on digital device
  To assess the effect of 84 days of IP consumption on severity of the symptoms using Computer Vision Syndrome-Questionnaire.The two levels of intensity, or strength of the symptom, will be graded similarly, on a scale of 1 to 2 points, where moderate = 1 and intense = 2. In the analysis, a symptom rated as never occurring will be treated as 0 (none) on the intensity scale.
  The overall assessment will be conducted by obtaining the total score for DES. The result of frequency X intensity will be recorded as: 0 = 0; 1 or 2 = 1; 4 = 2. If the total score is ≥ 6 points, the participant will be considered to be suffering from digital eye strain. It is further categorized as mild DES (score = 6-12), moderate DES (score = 13-18), and severe DES (score = 19-32)
Computer Vision Syndrome-Questionnaire | Day 28 before playing videogames on digital device
  To assess the effect of 84 days of IP consumption on severity of the symptoms using Computer Vision Syndrome-Questionnaire.The two levels of intensity, or strength of the symptom, will be graded similarly, on a scale of 1 to 2 points, where moderate = 1 and intense = 2. In the analysis, a symptom rated as never occurring will be treated as 0 (none) on the intensity scale.
  The overall assessment will be conducted by obtaining the total score for DES. The result of frequency X intensity will be recorded as: 0 = 0; 1 or 2 = 1; 4 = 2. If the total score is ≥ 6 points, the participant will be considered to be suffering from digital eye strain. It is further categorized as mild DES (score = 6-12), moderate DES (score = 13-18), and severe DES (score = 19-32)
Computer Vision Syndrome-Questionnaire | Day 56 before playing videogames on digital device
  To assess the effect of 84 days of IP consumption on severity of the symptoms using Computer Vision Syndrome-Questionnaire.The two levels of intensity, or strength of the symptom, will be graded similarly, on a scale of 1 to 2 points, where moderate = 1 and intense = 2. In the analysis, a symptom rated as never occurring will be treated as 0 (none) on the intensity scale.
  The overall assessment will be conducted by obtaining the total score for DES. The result of frequency X intensity will be recorded as: 0 = 0; 1 or 2 = 1; 4 = 2. If the total score is ≥ 6 points, the participant will be considered to be suffering from digital eye strain. It is further categorized as mild DES (score = 6-12), moderate DES (score = 13-18), and severe DES (score = 19-32)
Computer Vision Syndrome-Questionnaire | Day 84 before playing videogames on digital device
  To assess the effect of 84 days of IP consumption on severity of the symptoms using Computer Vision Syndrome-Questionnaire.The two levels of intensity, or strength of the symptom, will be graded similarly, on a scale of 1 to 2 points, where moderate = 1 and intense = 2. In the analysis, a symptom rated as never occurring will be treated as 0 (none) on the intensity scale.
  The overall assessment will be conducted by obtaining the total score for DES. The result of frequency X intensity will be recorded as: 0 = 0; 1 or 2 = 1; 4 = 2. If the total score is ≥ 6 points, the participant will be considered to be suffering from digital eye strain. It is further categorized as mild DES (score = 6-12), moderate DES (score = 13-18), and severe DES (score = 19-32)

SECONDARY OUTCOMES:
Asthenopia Visual Fatigue Likert scale | Day 0, day 14, day 28, day 56 and day 84.
  The participant will respond digitally a relevant present condition from None (0), Very Mild (1), Mild (2), Moderate (3), Very Moderate (4), and Severe (5) and the total score will be calculated
Immunitythe subject felt sick will be documented in sick diary along with the concomitant medication used (dose and frequency will be captured). | Day 14, Day 28, Day 56 and Day 84
  the number of days when the subject felt sick will be documented in sick diary along with the concomitant medication used (dose and frequency will be captured). Immunity as assessed by the number of sick days reported for each participant during the treatment period, as compared to the placebo
Immunity of participan has contracted the common cold/flu | Day 14, Day 28, Day 56 and Day 84
  Immunity as assessed by the number of times participant has contracted the common cold/flu during the treatment period, as compared to the placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Shalini Srivastava, MD medicine, Principal Investigator — Vedic Lifesciences Pvt. Ltd.
Locations (3):
- India (3):
  - Aman Hospital and Research Center, Ahmedabad, Guijarat
  - Wavikar Eye Institute, Thane, Maharashtra
  - Jaipur National University Institute for Medical Sciences & Research Centre, Jaipur, Rajasthan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hecht KA, Marwah M, Wood V, Nishida Y, Bach AE, Gerson J, Hom MM, Schnackenberg J, Raote S, Srivastava S, Negi P, Caston E. Astaxanthin (AstaReal(R)) Improved Acute and Chronic Digital Eye Strain in Children: A Randomized Double-Blind Placebo-Controlled Trial. Adv Ther. 2025 Apr;42(4):1811-1833. doi: 10.1007/s12325-025-03125-7. Epub 2025 Feb 27. PMID 40014233